CLINICAL TRIAL: NCT00488202
Title: Advanced Ovarian Cancer and Sexuality Phase 1
Acronym: ANOVA1
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Other Study IDs: H06-03235
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer; Sexual Function
Keywords: Advanced Ovarian Cancer; Sexual Function
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Women with Advanced Ovarian Cancer (AOC) suffer from severe sexual side effects from treatment. The prevalence of the sexual issues is not known.

The degree to which these sexual side effects is affected by treatment is also not known, as the literature in this area focuses on post-treatment analysis.

Specific Aim #1 (Quantitative Phase): To determine the prevalence and types of sexual difficulties using self-report questionnaires in women about to receive treatment for Stage III or IV Ovarian Cancer at the BCCA and over time, and to correlate these symptoms with degree of cancer symptoms, well-being, depressive symptoms, and relationship satisfaction

DETAILED DESCRIPTION:
Hypothesis 1a: Compared to baseline pre-treatment data, and to existing data for women with early-stage gynaecologic cancer, rates of sexual difficulties will be significantly higher and frequency of sexual intercourse will be significantly lower in women with advanced ovarian cancer. We hypothesize that difficulties specifically in the domains of sexual desire, sexual distress, and genital pain will be the most common types of sexual dysfunction to characterize women with advanced ovarian cancer.

Hypothesis 1b: We hypothesize that the degree of sexual symptoms will be significantly greater at 3 months and 10 months post-treatment than compared to pre-treatment, and that sexual difficulties may be significantly greater at 3 months post-treatment than at 10-months post-treatment.

Hypothesis 1c: We hypothesize that degree of sexual difficulty and sexual distress will be significantly correlated with (a) overall well-being; (b) depressive symptoms; and (c) relationship satisfaction.

Hypothesis 1d: As an exploratory analysis, we will investigate the relationship of ovarian cancer-related variables (i.e., type of treatment, duration of treatment, number of medications), and demographic variables (i.e., age, relationship duration, education) on each of the hypotheses in 1a - 1c.

ELIGIBILITY:
Inclusion Criteria:

* Women with Advanced Ovarian Cancer (AOC) who have not received treatment yet, but who are seeking treatment at the BC Cancer Agency.
* Women must be able to understand English enough to fill out the questionnaire packages.
* Mastery of written English is required. No translation services will be available for this study.

Exclusion Criteria:

* Anyone without an AOC diagnosis, who are not seeking treatment at BCCA, or who cannot understand enough English to complete the questionnaires will be excluded.
* Those who do not have a mastery of written English are excluded.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women diagnosed with advanced ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — UBC
Locations (2):
- Canada (2):
  - UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia
  - UBC Sexual Health Lab, Vancouver, British Columbia